CLINICAL TRIAL: NCT05532722
Title: A Study of ABC008 in Subjects with T-cell Large Granular Lymphocytic Leukemia (T-LGLL)
Brief Title: ABC008 in Subjects with T-cell Large Granular Lymphocytic Leukemia (T-LGLL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abcuro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABC008-LGL-101
Record Dates: First submitted 2022-08-19; First posted 2022-09-08 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: T-cell Large Granular Lymphocytic Leukemia
Keywords: T-cell Large Granular Lymphocytic Leukemia; T-LGLL
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- ABC008 Dose Level 1 Cohort (Experimental): 0.25 mg / kg ABC008 Subjects receive ABC008 every 8 weeks.
  Cohorts receive escalating doses of ABC008 until completion of cohort 5 or any cohort is determined to have exceeded the maximum tolerated dose.
  Interventions: Drug: ABC008
- ABC008 Dose Level 2 Cohort (Experimental): 0.75 mg / kg ABC008 Subjects receive ABC008 every 8 weeks.
  Cohorts receive escalating doses of ABC008 until completion of cohort 5 or any cohort is determined to have exceeded the maximum tolerated dose.
  Interventions: Drug: ABC008
- ABC008 Dose Level 3 Cohort (Experimental): 1.5 mg / kg ABC008 Subjects receive ABC008 every 8 weeks.
  Cohorts receive escalating doses of ABC008 until completion of cohort 5 or any cohort is determined to have exceeded the maximum tolerated dose.
  Interventions: Drug: ABC008
- ABC008 Dose Level 4 Cohort (Experimental): 3.0 mg / kg ABC008 Subjects receive ABC008 every 8 weeks OR 1.5 mg / kg Subjects receive ABC008 every 4 weeks.
  Cohorts receive escalating doses of ABC008 until completion of cohort 5 or any cohort is determined to have exceeded the maximum tolerated dose.
  Interventions: Drug: ABC008
- ABC008 Dose Level 5 Cohort (Experimental): 3.0 mg / kg ABC008 Subjects receive ABC008 every 4 weeks.
  Cohorts receive escalating doses of ABC008 until completion of cohort 5 or any cohort is determined to have exceeded the maximum tolerated dose.
  Interventions: Drug: ABC008

INTERVENTIONS:
Drug: ABC008 — Given subcutaneous injection

SUMMARY:
An open label, ascending dose study for adult subjects with T-cell Large Granular Lymphocytic Leukemia (T-LGLL)

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age.
* Has body mass index (BMI) ≤35 kg/m2.
* Has a documented diagnosis of T LGLL.
* Has any 1 or more of the following at Screening:

  * Absolute neutrophil count (ANC) <0.5 x 109/L
  * ANC ≥0.5 x 109/L and <1.0 x 109/L associated with recurrent infection (≥2 or more infections requiring antimicrobial therapy within the previous 12 months)
  * Hemoglobin (Hgb) <8 g/dL or packed red blood cell transfusion frequency ≥1 time in the 4 weeks immediately prior to Screening
  * Hgb ≥8 g/dL and <10 g/dL accompanied by documented symptoms of anemia, e.g., fatigue, weakness, pale or yellowish skin, irregular heartbeat, shortness of breath, dizziness, or lightheadedness.
* Has adequate hepatic and renal function at Screening, as indicated by:

  * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST); <2.5x the upper limit of normal (ULN)
  * Total bilirubin ≤1.5 ULN; subjects with Gilbert syndrome must have a total bilirubin <3.0x ULN with direct bilirubin <1.0x ULN at time of Screening
  * Estimated glomerular filtration rate (eGFR) ≥45 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation corrected for the body surface area of the subject calculated by the Mosteller equation and divided by 1.73
* Agrees to adhere to the current Centers for Disease Control advice regarding minimizing exposure to severe acute respiratory syndrome coronavirus 2 (SARS CoV 2) from the first Screening Visit until the End of Study (EOS)/Early Termination Visit (ETV).

Exclusion Criteria:

* Has reactive large granular lymphocytosis.
* Has active anemia secondary to confirmed etiologies other than T-LGLL, including known vitamin or mineral deficiency, gastrointestinal bleeding, or genetic disorder; or has active neutropenia secondary to known vitamin or mineral deficiencies or genetic disorder.
* Has a platelet count ≤20 x 109/L or other clinically significantly abnormal laboratory results not related to the underlying condition in the Investigator's or Sponsor's opinion at Screening.
* Has known hypersensitivity to any component of the formulation of ABC008, or history of anaphylaxis to any prior mAb therapy.
* Has any other autoimmune or autoinflammatory disease other than RA, inclusion body myositis (IBM), secondary Sjogren's syndrome (SS), or thyroid disease.
* Has another myelo /lympho proliferative disorder or malignancy (other than monoclonal gammopathy of unknown significance [MGUS] not requiring treatment) within the past 5 years prior to Screening except completely resected nonmelanoma skin cancer, curatively treated localized prostate cancer, and completely resected carcinoma in situ at any site.
* Has a current diagnosis of active tuberculosis (TB)
* Has a history of herpes zoster infection that was disseminated, required hospitalization, or IV antiviral therapy in the 24 weeks prior to Day 1.
* Active, chronic, or past history of hepatitis B virus or hepatitis C virus (HCV) infection (hepatitis B core antibody or surface antigen positive, or HCV antibody positive with reflex HCV ribonucleic acid [RNA] positive at Screening; individuals who have received curative therapy for HCV are permitted if therapy was completed at least 24 weeks prior to Screening and subject is HCV RNA negative);
* Has known active bacterial, viral, fungal, or atypical mycobacterial infection, or any major episode of infection that required hospitalization
* Has received live (including attenuated) vaccination in the 30 days prior to Day 1 or killed vaccine within 14 days prior to Day 1.
* Is human immunodeficiency virus (HIV) positive by antigen/antibody test, human T cell lymphotropic virus (HTLV 1 or 2) positive by antibody test.
* Has had major surgery (defined as surgery requiring general or regional anesthesia) within 6 weeks prior to Day 1 or is expected to receive surgery during the study.
* Has a history of organ transplant (e.g., solid, bone marrow) or is expected to receive one during the study.
* Has any other condition or social situations that would interfere with the subject's study participation, increase the risk associated with study participation or investigational product administration, interfere with the interpretation of study results, or would otherwise make the subject inappropriate for entry into this study in the Investigator's or Sponsor's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of treatment-emergent AEs and SAEs as determined by NCI CTCAE v5.0 | Through Study Completion an average of 48 weeks

SECONDARY OUTCOMES:
Change from baseline in safety lab (Hematology) | Through Study Completion an average of 48 weeks
Change from baseline in safety lab (Chemistry) | Through Study Completion an average of 48 weeks
Change from baseline in safety lab (Coagulation) | Through Study Completion an average of 48 weeks
  Includes the following coagulation labs: INR and aPTT
Change from baseline in safety lab (Complement) | Through Study Completion an average of 48 weeks
  Includes the following complement labs: C3 and CH50
Change from baseline in safety lab (Cytokines) | Through Study Completion an average of 48 weeks
Change from baseline in safety lab (CMV Viral Load) | Through Study Completion an average of 48 weeks
Change from baseline in safety lab (EBV Viral Load) | Through Study Completion an average of 48 weeks
Change from baseline in ECG (Rhythm) | Through Study Completion an average of 48 weeks
Change from baseline in ECG (Heart Rate) | Through Study Completion an average of 48 weeks
Change from baseline in ECG parameters | Through Study Completion an average of 48 weeks
  Includes the following ECG parameters: RR interval, PR interval, QRS interval, QT interval, QT interval corrected by Bazett's formula, and QTcF
Change from baseline in vital sign (Systolic and diastolic blood pressure) | Through Study Completion an average of 48 weeks
Change from baseline in vital sign (temperature) | Through Study Completion an average of 48 weeks
Change from baseline in vital sign (respiratory rate) | Through Study Completion an average of 48 weeks
Change from baseline in vital sign (pulse rate) | Through Study Completion an average of 48 weeks
Percentage of subjects demonstrating overall response (defined as total number of subjects with CR or PR) at all time points assessed | Day 1 and throughout the 48 weeks of follow up
Percentage of subjects demonstrating complete response at all time points assessed | Day 1 and throughout the 48 weeks of follow up
  A complete response is defined by normalization of hemoglobin, neutrophil and platelet levels without transfusion
Percentage of subjects demonstrating partial response at all time points assessed | Day 1 and throughout the 48 weeks of follow up
  A partial response is defined by improvement in any of the following criteria but not all: hemoglobin, neutrophil and platelet levels without transfusion
Duration of response at all time points assessed | Day 1 and throughout the 48 weeks of follow up
Overall survival at Week 48 | Day 1 and throughout the 48 weeks of follow up
The change from baseline in levels of KLRG1 expressing lymphocytes over time | Day 1 and throughout the 48 weeks of follow up
The change from baseline in levels of T-LGL counts over time | Day 1 and throughout the 48 weeks of follow up
The change from baseline in levels of lymphocyte subsets over time | Day 1 and throughout the 48 weeks of follow up
The maximum serum concentration [CMax] of ABC008 | Day 1 and throughout the 48 weeks of follow up
The time to maximum concentration [TMax] of ABC008 | Day 1 and throughout the 48 weeks of follow up
The area under the concentration-time curve [AUC] of ABC008 | Day 1 and throughout the 48 weeks of follow up
The apparent clearance [CL/F] of ABC008 | Day 1 and throughout the 48 weeks of follow up
The apparent volume of distribution [Vd/F] of ABC008 | Day 1 and throughout the 48 weeks of follow up
The elimination half-life [t½] of ABC008 | Day 1 and throughout the 48 weeks of follow up

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - University of Southern California, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided